CLINICAL TRIAL: NCT02493140
Title: Evaluation of Efficacy and Safety of a Cashew Apple Extract on Weight Management and Associated Metabolic Risk Factors in Overweight/Obese Volunteers: a Randomized, Double-blind, Placebo-controlled, Parallel-group Clinical Trial
Brief Title: Evaluation of Efficacy of a Cashew Apple Extract on Weight Management and Associated Metabolic Risk Factors in Overweight/Obese Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dialpha (Other)
Collaborators: Naturalpha (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2015-A00160-49
Record Dates: First submitted 2015-07-06; First posted 2015-07-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Weight Loss
Keywords: Weight management; cashew apple extract; overweight
MeSH Terms: conditions — Weight Loss; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cashew apple extract (Cashewin) (Active Comparator)
  Interventions: Dietary Supplement: Cashew apple extract (Cashewin)
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cashew apple extract (Cashewin) — 6 capsules per day (2 capsules 3 times per day, to be taken before breakfast, lunch and diner, each capsule containing 200 mg of Cashewin) during 12 weeks
  Arms: Cashew apple extract (Cashewin)
Dietary Supplement: Placebo — 6 capsules per day (2 capsules 3 times per day, to be taken before breakfast, lunch and diner) during 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of a cashew apple extract on weight management and associated metabolic risk factors in overweight/obese volunteers, versus placebo, after 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* 27 ≤ BMI ≤ 35 kg/m²
* Abdominal obesity
* Acceptance to adhere to diet and physical activity recommendations while maintaining global lifestyle habits
* Stable body weight (<5% variation) within the last 3 months prior to screening

Exclusion Criteria:

* Allergy to nuts and products thereof and allergy to mango fruit
* Type I or II diabetes
* Smokers
* Severe chronic diseases
* History of bariatric surgery and eating disorders
* Use of weight management products or medications which could affect nutrients absorption, lipids or carbohydrates metabolism

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2015-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Body weight reduction | 12 weeks

SECONDARY OUTCOMES:
Body weight variation | 6 weeks and 12 weeks
Body fat variation | 6 and 12 weeks
BMI variation | 6 and 12 weeks
Waist and hip circumferences variation | 6 and 12 weeks
Fasting glycemia variation | 12 weeks
Fasting insulinemia variation | 12 weeks
HOMA-IR index variation | 12 weeks
Variation of glycemia 2h post glucose solution intake | 12 weeks
Blood lipids (total cholesterol, HDL, LDL, triglycérides) variation | 12 weeks
CRPus variation | 12 weeks
Systolic and diastolic blood pressure variation | 6 and 12 weeks
Safety (blood parameters measurements: urea, creatinine, ASAT, ALAT) with adverse events recording | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Deplanque, Principal Investigator — Naturalpha
Locations (1):
- Clinical Nutrition Center Naturalpha (CNCN), Lille, France

REFERENCES:
- [Background] Janssen I, Katzmarzyk PT, Ross R. Waist circumference and not body mass index explains obesity-related health risk. Am J Clin Nutr. 2004 Mar;79(3):379-84. doi: 10.1093/ajcn/79.3.379. PMID 14985210
- [Background] Ribeiro da Silva LM, Teixeira de Figueiredo EA, Silva Ricardo NM, Pinto Vieira IG, Wilane de Figueiredo R, Brasil IM, Gomes CL. Quantification of bioactive compounds in pulps and by-products of tropical fruits from Brazil. Food Chem. 2014 Jan 15;143:398-404. doi: 10.1016/j.foodchem.2013.08.001. Epub 2013 Aug 9. PMID 24054258
- [Background] Kuczmarski RJ, Flegal KM. Criteria for definition of overweight in transition: background and recommendations for the United States. Am J Clin Nutr. 2000 Nov;72(5):1074-81. doi: 10.1093/ajcn/72.5.1074. PMID 11063431
- [Background] P. Suganya and R. Dharshini. Value added products from cashew apple - an alternate nutritional source. International Journal of current research, Vol. 3, Issue 7, pp. 177-180, July 2011
- [Background] Prasertsri P, Roengrit T, Kanpetta Y, Tong-Un T, Muchimapura S, Wattanathorn J, Leelayuwat N. Cashew apple juice supplementation enhanced fat utilization during high-intensity exercise in trained and untrained men. J Int Soc Sports Nutr. 2013 Mar 7;10(1):13. doi: 10.1186/1550-2783-10-13. PMID 23497120
- [Background] Vergara CMAC, Honorato TL, Maia GA, Rodrigues S. Prebiotic effect of fermented cashew apple (Anacardium occidentale L) juice. LWT-Food Sci Technol. 2010; 43:141-145.
- See also: Identification, Evaluation and Treatment of Overweight and Obesity in Adults — http://www.nhlbi.nih.gov/files/docs/guidelines/prctgd_c.pdf
- See also: Clinical guidelines on the Identification, Evaluation, and Treatment of Overweight and Obesity in adults — http://www.nhlbi.nih.gov/files/docs/guidelines/ob_gdlns.pdf